CLINICAL TRIAL: NCT02375360
Title: Quality of Life in Food Allergic Patients Before, During and After Oral Immunotherapy
Brief Title: OIT Effect on FAQLQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 52/14
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (7):
- Children 8-12- control: Children aged 8-12 years with food allergy who are not undergoing oral immunoterapy
- Parents 0-12 - control: Parents to children aged 0-12 years with food allergy who are not undergoing oral immunoterapy
- Children 8-12 - OIT: Children aged 8-12 years with food allergy who are undergoing oral immunoterapy
  Interventions: Other: Oral immunotherapy
- Teenagers 13-17 - OIT: Teenagers aged 13-17 years with food allergy who are undergoing oral immunoterapy
  Interventions: Other: Oral immunotherapy
- Adults >18 - OIT: Adults> 18 years with food allergy who are undergoing oral immunoterapy
  Interventions: Other: Oral immunotherapy
- Parents 0-12 - OIT: Parents to children aged 0-12 years with food allergy who are undergoing oral immunoterapy
  Interventions: Other: Oral immunotherapy
- Parents 13-17 - OIT: Parents to teenagers aged 13-17 years with food allergy who are undergoing oral immunoterapy
  Interventions: Other: Oral immunotherapy

INTERVENTIONS:
Other: Oral immunotherapy
  Groups: Adults >18 - OIT; Children 8-12 - OIT; Parents 0-12 - OIT; Parents 13-17 - OIT; Teenagers 13-17 - OIT

SUMMARY:
Patients with food allergy and their parents will answer a food allergy quality of life questionnaire that will be translated to Hebrew and validated. Questionnaires will be filled also by patients undergoing oral immunotherapy (OIT).

DETAILED DESCRIPTION:
The food allergy quality of life questionnaires (FAQLQ) for children 8-12 y/o, teenagers 13-17 y/o and adults > 18 y/o and parents to children 0-12 y/o and to teenagers will be translated to Hebrew. Questionnaires will be given to patients with food allergy followed at Asaf Harofeh Medical Center. Questionnaires will be examined for internal consistency. The Food Allergy Independent Measure (FAIM) questionnaire for the same age groups will also be translated to Hebrew. The FAQLQ will be validated by correlation with the FAIM.

The questionnaires will then be administered to patients and families undergoing food oral immunotherpy, before during and following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected food allergy

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children, teenagers and their parents and adults with food allergy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 1 - 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Harofeh Medical Center, Ẕerifin, Israel, Israel